CLINICAL TRIAL: NCT02724085
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single-Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenous TP-271 in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Assess the Safety, Tolerability and PK of IV TP-271
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TP-271-001; HHSN272201100028C (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2015-09-04; First posted 2016-03-31 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — TP-271

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 0.15 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort B (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 0.45 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort C (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 1.0 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort D (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 2.0 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort E (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 3.0 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort F (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 4.0 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271
- Cohort G (Active Comparator): IV dose of TP-271, a novel, broad-spectrum tetracycline-class antibiotic, 5.0 mg/kg single dose, 60 minute infusion or Placebo - sterile 0.45% saline for 60 minute IV infusion
  Interventions: Drug: TP-271

INTERVENTIONS:
Drug: TP-271 — TP-271 is a novel, broad-spectrum tetracycline with potent activity against multidrug-resistant pathogens. It will be administered intravenously (IV) in doses ranging from 0.15 to 5.0 mg/kg

SUMMARY:
This is a single-center, randomized, placebo-controlled, double-blind, single-ascending-dose, inpatient study to assess the safety, tolerability, and pharmacokinetics of TP-271 in healthy subjects. Subjects aged 18 to 50 years who fulfill the inclusion/exclusion criteria will be enrolled in this study.

DETAILED DESCRIPTION:
Up to seven cohorts of eight subjects each (up to a total of 56 subjects) will be enrolled. The eight subjects within each cohort will be randomized 6:2 to receive a single intravenous dose of TP-271 or placebo. The planned doses are:

Cohort A: 0.15 mg/kg Cohort B: 0.45 mg/kg Cohort C: 1.0 mg/kg Cohort D: 2.0 mg/kg Cohort E: 3.0 mg/kg Cohort F: 4.0 mg/kg Cohort G: 5.0 mg/kg

Doses of IMP will be administered intravenously on the morning of Day 1 following an overnight fast (minimum 8 hours).

During the Screening Period (within the 28 days prior to the subject receiving TP-271 or placebo) each subject will be assessed for eligibility. Each subject must sign and date an ICF prior to undergoing any study-related procedures.

All cohorts will follow the same study design (Figure 1). On Day -1, subjects will be admitted to the study unit so their eligibility can be confirmed. Subjects will be required to stay overnight at the study unit on Day -1. On Day 1, eligible subjects will be enrolled and randomized to receive either TP-271 or placebo. Subjects will be required to stay at the study unit from Day 1 through Day 5 to assess safety and obtain required PK samples. On Day 5, subjects will be discharged from the study unit. A final safety assessment will be performed once between Day 7 and Day 10 following the subject's dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Be within the age range of 18 to 50 years, inclusive, at the time of Screening.
2. Voluntarily sign an IRB/Research Ethics Committee (IRB/REC)-approved ICF to participate in the study after all relevant aspects of the study have been explained and discussed with the subject and before undergoing any study related procedures.
3. Have a body mass index (BMI) ≥18.0 and ≤33.0 kg/m2.
4. Be clear of any history of, and have negative screen for, HIV 1 and 2 and hepatitis B and C.
5. Have the ability to communicate with the investigative site staff in a manner sufficient to carry out all protocol procedures as described.
6. Females must be of non-child bearing potential, either 1-year post-menopausal or surgically sterile (bilateral oophorectomy, bilateral tubal ligation, or complete hysterectomy).
7. Male subjects must be willing and able to use a barrier method of birth control or practice abstinence (even if they have had a vasectomy) from dosing through 90 days after the dose of IMP.

Exclusion Criteria:

1. History and/or presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal, and psychiatric/mental disease/disorders, which, in the opinion of the PI, may either put the subject at risk because of participation in the study, influence the results of the study, or influence the subject's ability to participate in the study.
2. Clinical laboratory values that fall outside the eligibility range specified in the table in Appendix C are exclusionary. For the laboratory values that are not included in Appendix C, values outside of the reference range are exclusionary with the following exceptions:

   Low Chemistry Values High Chemistry Values Out of Range UA Out of Range Hematology Bicarbonate (> 18 mEq/L Chloride GGT HDL Cholesterol LDH LDL Cholesterol Phosphorus Triglycerides Chloride HDL Cholesterol LDL Cholesterol Phosphorus Triglycerides High or low specific gravity Cloudy Mucus Crystals Ketones (when blood glucose is normal) Hyaline casts High or low pH

   High hematocrit Basophils Monocytes MCV MCHC MCH RBC
3. Blood pressure and pulse outside of the following ranges are exclusionary:

   * Systolic blood pressure 85 - 145 mm Hg
   * Diastolic blood pressure 50 - 95 mm Hg
   * Pulse rate 45 - 95 beats per minute (bpm)
4. Known allergy to tetracycline antibiotics or to any of the excipients in TP-271.
5. Clinically significant abnormal 12-lead ECG, including the following:

   * Rhythm other than sinus, QTc interval using Fridericia's formula (QTcF) >450 msec;
   * Evidence of second- or third-degree atrioventricular (AV) block;
   * Pathological Q-waves (defined as Q-wave >40 msec or depth >0.4 to 0.5 mV);
   * Evidence of ventricular pre-excitation;
   * Electrocardiographic evidence of complete left bundle branch block, right bundle branch block (RBBB), incomplete LBBB;
   * Intraventricular conduction delay with QRS duration >120 msec;
   * ST segment abnormalities unless judged by the Investigator to be non-pathologic.
6. History of seizures.
7. A history within 3 years of Screening of drug abuse (including benzodiazepines, opioids, amphetamine, and cocaine) or a positive drug result at Screening for any of these drugs of abuse. Also excluded are subjects who test positive for cannabinoids (THCs).
8. Use of tobacco, nicotine, or nicotine-replacement products within the 3 months prior to the dose of study drug through the last study visit.
9. Typical weekly alcohol consumption of 7 or more alcoholic drinks. One drink is defined as 1 glass of beer (approximately 10 to 12 oz) or 1 can (12 oz) of beer, 1 glass of wine (approximately 4 to 5 oz), or 1 glass of distilled spirits (hard liquor) containing 1 oz of the liquor (1 oz of liquid is approximately 30 mL).
10. Alcohol consumption within 48 hours prior to dosing.
11. Participation in a clinical trial within 10 half-lives of the prior study treatment or the past 3 months if the half-life is unknown of dose or planned participation in another trial in addition to this one during the trial.
12. History of difficulty in donating blood or poor venous access.
13. Subject has donated blood (1 unit or 350 mL) within 1 month prior to receiving test material or plans to donate prior to receiving test material or during the trial.
14. Use of any prescription or non-prescription medication, including vitamins or herbal medications, within 7 days, or 5 half-lives (if known), whichever is longer, prior to dosing. The use of acetaminophen, naproxen, and ibuprofen is permitted except for within 24 hours prior to dosing. (Note: Subjects must refrain from taking herbal or dietary supplements or prescription drug therapy for the duration of the study.)
15. Unwillingness or inability to follow the procedures outlined in the protocol. Subject is mentally or legally incapacitated

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Through study completion, appromiximately 39 days
  The incidence, intensity, and type of adverse events (AE)
  Outcome measures to be collected in support of the primary objective (safety and tolerability) include:
  * The incidence, intensity, and type of AEs (from time of signing of informed consent form [ICF] through EOS);
  * Changes in physical examination findings (Day -1 and EOS);
  * Changes in vital signs (Day -1 through EOS);
  * Changes in safety laboratory (chemistry, hematology, coagulation, urinalysis) results (Days -1 through EOS); and
  * Changes in ECG measurements (Days -1 through EOS).
Physical Exams | Through study completion, appromiximately 39 days
  Changes in physical examination findings
Vital Signs | Through study completion, appromiximately 39 days
  Changes in vital signs
Safety Laboratory | Through study completion, appromiximately 39 days
  Changes in safety laboratory (chemistry, hematology, coagulation, urinalysis) results
ECG measurements | Through study completion, appromiximately 39 days
  Changes in ECG measurements

SECONDARY OUTCOMES:
Plasma Pharmacokinetic (PK) Analysis | Days 1-5
  Plasma concentrations of TP-271 and its C-4 epimer TP-9555 for PK analysis
Urine Pharmacokinetic (PK) Analysis | Days 1-5
  Urine concentrations of TP-271 and its C-4 epimer TP-9555
PK parameters - Cmax | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Cmax [The maximum observed plasma concentration]
PK parameters - Tmax | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Tmax [The time from dosing at which Cmax is apparent]
PK parameters - C8 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C8 [The concentration at 8 hours post-dose]
PK parameters - C12 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C12 [The concentration at 12 hours post-dose]
PK parameters - C24 | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for C24 [The concentration at 24 hours post-dose]
PK parameters - AUC(0-last) | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC(0-last) [The area under the concentration vs time curve from zero to the last measured time point]
PK parameters - AUC(0-inf) | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC(0-inf) [The area under the concentration vs time curve from time zero extrapolated to infinity]
PK parameters - AUC%extrap | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for AUC%extrap [The percentage of AUC(0-inf) accounted for by extrapolation]
PK parameters - Lambda-z | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Lambda-z [Slope of the regression line passing through the apparent elimination phase in a concentration vs time plot]
PK parameters - T1/2el | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for T1/2el [The elimination half-life]
PK parameters - CL | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for CL [Clearance: the volume of plasma cleared per unit time]
PK parameters - Vd | Days 1-5
  PK parameters will be calculated from the plasma concentration versus time data (as appropriate) for Vd [The volume of distribution]
PK parameters - epimer/parent | Days 1-5
  The PK parameters of the epimer/parent will be calculated for Cmax and AUC(0-inf).

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided